CLINICAL TRIAL: NCT00879944
Title: Impact of the Severity of Pediatric Psoriasis on Childhood Body Mass Index and Comorbid Risk Factors: an Epidemiologic Analysis
Brief Title: Impact of the Severity of Pediatric Psoriasis on Childhood Body Mass Index
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Amy Paller, Chair, Department of Dermatology, Professor of Dermatology and Pediatric Dermatology, Northwestern University
Other Study IDs: AP-2009-13793
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Psoriasis; Atopic Dermatitis
Keywords: Psoriasis; Obesity; BMI; Atopic Dermatitis
MeSH Terms: conditions — Psoriasis; Dermatitis, Atopic; Obesity | interventions — Blood Pressure; Body Height; Weights and Measures; Waist Circumference

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Psoriasis: Children ages 5-17 years old with moderate or severe plaque type psoriasis. Blood pressure will be measured once while patient is seated Height will be measured in centimeters at the time of enrollment Weight will be measured in kilograms at enrollment Body Mass Index (BMI) will be calculated from a subject's height and weight Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest with an inelastic measuring tape at the end of normal expiration to the nearest 0.1cm
  Interventions: Other: Blood pressure; Other: Height; Other: Weight; Other: BMI; Other: Waist Circumference
- Atopic Dermatitis Controls: Children ages 5 to 17 years old with moderate to severe atopic dermatitis. Blood pressure will be measured once while patient is seated Height will be measured in centimeters at the time of enrollment Weight will be measured in kilograms at enrollment Body Mass Index (BMI) will be calculated from a subject's height and weight Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest with an inelastic measuring tape at the end of normal expiration to the nearest 0.1cm
  Interventions: Other: Blood pressure; Other: Height; Other: Weight; Other: BMI; Other: Waist Circumference
- Healthy Controls: Children 5-17 years of age who are healthy and seen in dermatology clinic for a non-systemic skin condition.
  Blood pressure will be measured once while patient is seated Height will be measured in centimeters at the time of enrollment Weight will be measured in kilograms at enrollment Body Mass Index (BMI) will be calculated from a subject's height and weight Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest with an inelastic measuring tape at the end of normal expiration to the nearest 0.1cm
  Interventions: Other: Blood pressure; Other: Height; Other: Weight; Other: BMI; Other: Waist Circumference

INTERVENTIONS:
Other: Blood pressure — Blood pressure will be measured once while patient is seated
Other: Height — Height will be measured in centimeters at the time of enrollment
Other: Weight — Weight will be measured in kilograms at enrollment
Other: BMI — Body Mass Index (BMI) will be calculated from a subject's height and weight
Other: Waist Circumference — Waist circumference will be measured midway between the lowest rib and the superior border of the iliac crest with an inelastic measuring tape at the end of normal expiration to the nearest 0.1cm

SUMMARY:
The object of this research study is to examine these associations in children as very little is known about psoriasis and cardiovascular risk factors in the pediatric population.

DETAILED DESCRIPTION:
Several environmental factors and comorbid conditions have been found to be associated with psoriasis in adults, including obesity, depression, smoking, and other cardiovascular risk factors such as high blood pressure. The object of this research study is to examine these associations in children as very little is known about psoriasis and cardiovascular risk factors in the pediatric population.

This is a multi-center study with a planned total enrollment of about 200 subjects ages 2-17 years old with psoriasis and 100 aged-match controls. Patient and family history will be recorded. All subjects will undergo standard height, weight, blood pressure, and waist circumference (WC). For the obese and overweight subjects we will also obtain their growth charts to attempt to correlate weight gain with psoriasis onset and progression. All data will be compiled and then statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be between the ages of 5 and 17 years at the time of enrollment.
* Subjects of either sex.
* Subjects who have had psoriatic plaques for more than 6 months.
* Subjects and guardians of minors must sign the approved IRB consent form(s) prior to initiation of the study protocol.
* Subjects enrolled as "non-inflammatory" normal controls will carry a common non- systemic skin condition, such as acne, nevi, warts and molluscum as their main diagnosis.
* Subjects enrolled as "inflammatory" normal controls will carry a diagnosis of moderate to severe atopic dermatitis.

Exclusion Criteria:

* Subjects who are unable to give informed consent or assent.
* Subjects who have had psoriasis for less than 6 months.
* Subjects whose condition is deemed unsafe or incapable by the study investigator for study participation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 1. Children ages 5 to 17 years old with either moderate or severe plaque type psoriasis
  2. Children ages 5 to 17 years old with moderate or severe atopic dermatitis
  3. Children ages 5 to 17 years old seen in dermatology clinic who are healthy and without a systemic disorder.
Sampling Method: Probability Sample
Enrollment: 409 (Actual)
Dates: Start 2009-05; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
BMI | 07/2010

SECONDARY OUTCOMES:
Blood Pressure | 07/2010
Waist circumference | 07/2010

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Paller, MD, Principal Investigator — Northwestern University
Locations (14):
- United States (9):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University School of Medicine, Stanford, California
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - UMass Memorial Dermatology Center, Worcester, Massachusetts
  - Central Dermatology, St Louis, Missouri
  - University Hospitals, Case Medical Centers, Cleveland, Ohio
  - Texas Dermatology Associates, Dallas, Texas
  - Texas Children's Hospital, Houston, Texas
- Nexus Clinical Resarch, St. John's, Newfoundland and Labrador, Canada
- Pontificia Universidad Catolica de Chile, Santiago, Chile
- University of Hong Kong, Tuenmen, Hong Kong
- Universita Verona, Verona, Italy
- UMC St. Radboud, Nijmegen, Netherlands

REFERENCES:
- [Result] Paller AS, Mercy K, Kwasny MJ, Choon SE, Cordoro KM, Girolomoni G, Menter A, Tom WL, Mahoney AM, Oostveen AM, Seyger MM. Association of pediatric psoriasis severity with excess and central adiposity: an international cross-sectional study. JAMA Dermatol. 2013 Feb;149(2):166-76. doi: 10.1001/jamadermatol.2013.1078. PMID 23560297
- See also: Northwestern University Featured Clinical Trials Page — http://www.feinberg.northwestern.edu/depts/dermatology/research/clinical-trials/ctu-active%20trials.htm